CLINICAL TRIAL: NCT04496947
Title: Pilot Study Evaluating the Impact of Stress Reduction on Atherosclerotic : Heart and Mind Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Tawakol, Director, Nuclear Cardiology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2017P000706
Record Dates: First submitted 2020-07-29; First posted 2020-08-04 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-11

CONDITIONS: Atherosclerosis; Stress; Inflammation
MeSH Terms: conditions — Atherosclerosis; Inflammation | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: 2 groups:
  1. stress reduction intervention
  2. no intervention
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress Reduction (Experimental): 8 week stress reduction course
  Interventions: Behavioral: Stress Reduction
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Stress Reduction — The stress reduction program is a multimodal mind-body resiliency program that incorporates 3 core components into each session:
  * Elicitation of the Relaxation Response (RR) through mind-body techniques;
  * Discussion about stress awareness to learn how to identify personal stressors and experiences of stress; and
  * Coping strategies and adaptive perspective-taking to promote positive well-being.
  Arms: Stress Reduction

SUMMARY:
The plot study aims to evaluate the effect of 8 weeks of stress reducing intervention on atherosclerotic plaque inflammation in adults, as quantified by positron emission tomography (PET) with fluorine-2-deoxy-D-glucose (FDG) in individuals with increased psychosocial stress.

DETAILED DESCRIPTION:
This randomized controlled imaging study will be performed to evaluate the impact of mindfulness-based stress reduction via a mind body program on arterial inflammation in individuals with self-identified high levels of stress. Individuals will undergo baseline Fluorodeoxyglucose-Positron emission tomography / magnetic resonance imaging and will then be randomized to the stress-reduction intervention group or no intervention groups by blocks of 2:1, with stratification by age and sex. The stress reduction sessions focus on developing an understanding of stress physiology and the physiology of the relaxation response, on developing a regular practice of eliciting the relaxation response, and on learning cognitive behavioral and positive psychology/resilience skills.

During the screening period, patient acceptability for the study will be assessed based on medical history, concomitant medications, physical examination, and clinical laboratory test results. Acceptability for study participation will be confirmed for subjects who identify as having increased levels of stress and/or a Perceived Stress Scale score >5. Once the patient has passed screening, they will undergo baseline imaging followed by randomization and group assignment. Approximately 12 weeks after randomization, all individuals will return for follow-up imaging and evaluation.

Thus, 2 Fluorodeoxyglucose-Positron emission tomography / magnetic resonance imaging scans will be performed throughout the study for baseline and follow up to assess the intervention's impact on the brain and arterial inflammation, along with changes in related positron emission tomography / magnetic resonance imaging imaging parameters. Perceived Stress Scale will be delivered prior to Fluorodeoxyglucose-Positron emission tomography / magnetic resonance imaging, during both imaging visits to measure perceived psychological stress. During both imaging sessions, subjects will be exposed to overt faces to measure signals during brain imaging.

ELIGIBILITY:
Inclusion Criteria:

* • Aged between 30-65 years

  * Identifies as having increased levels of stress and/or has a Perceived Stress Scale (PSS) score >5 at baseline, and is interested in participating

Exclusion Criteria:

* Perceived Stress Scale (PSS) score <6

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in arterial inflammation by PET | 2 months
  Change in arterial inflammation based on FDG PET - from initial imaging to repeat imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Tawakol, MD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided